CLINICAL TRIAL: NCT05243901
Title: EPIPAGE2 Cohort Study Follow up at Ten and a Half Years
Brief Title: EPIPAGE 2 - 10-year Follow-up (RECONAI PROJECT)
Acronym: EPIPAGE2
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-68
Record Dates: First submitted 2022-02-02; First posted 2022-02-17 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Pre-Term; Development, Child
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Epipage 2 (Epidemiological study on small gestational ages) is a prospective population-based national cohort implemented to better understand the short, mid and long term future of premature children.

This study was launched on 28 March 2011 by the researchers of the EPOPé team (Perinatal, Obstetric and Pediatric Epidemiology Research) of the Epidemiology and Biostatistics Research Centre (INSERM U1153), in collaboration with the Inserm 1027 Unit (Epidemiology and Analysis in Public Health: risks, chronic diseases and handicaps) and medical teams of public health and research in 25 French regions.

The study focuses on children born before 35 weeks of amenorrhea.

3 follow-up steps for children included in the cohort have already been completed at 1, 2 and 5 and a half years of age. Currently, nearly 4,000 children are still eligible for follow-up.

Since the children are 9 years old, the follow-up steps are shared with those set up in another birth cohort, the Elfe cohort (Étude Longitudinale Française depuis l'Enfance, (www.elfe-france.fr) ), as part of the RE-CO-NAI project.

The RE-CO-NAI project is a research platform on cohorts of children followed since birth in order to be able to study in a global and multidisciplinary way the major issues of the health, development and socialization of children.

This RE-CO-NAI project was funded by the EQUIPEX 2011 call for projects as part of future investments.

This protocol, which is part of the RECONAI project, concerns the fully shared follow-up phase, proposed in the 10th year for the children of the two cohorts.

DETAILED DESCRIPTION:
The objectives of this new follow-up phase are to study:

* the relationships between prematurity, early growth and cardiometabolic disorders
* the relationship between parenting educational skills and children's quality of life
* the factors influencing children's puberty development
* the factors influencing the child's fitness and motor skills

Study design:

The 10 and a half year follow-up phase is a Category 2 Human Person Research (IHRP 2).

Study population The study population corresponds to all children who have participated in the Epipage 2 cohort since birth and whose parents did not wish to stop follow-up in the study. In total, nearly 4,000 children will be invited to participate in this new follow-up phase.

Methodology:

This follow-up phase will take place in 3 steps:

1. A telephone interview with one of the parents living regularly with the child. Parents will be asked to answer several questions concerning their family situation, the school (homework, school support), the health, sleep and nutrition of the child, the general health and mental health of the parent interviewed, the employment situation, the living conditions and educational practices of the family.
2. The home visit of the families of an investigator who will propose to the families several activities:

   * An interview with the child about his relations with his siblings, his comrades, his involvement in domestic activities and an estimate of his quality of life;
   * A physical examination measuring some of the child's health parameters and including tests of physical fitness and motor skills;
   * A test of the child's cognitive abilities;
   * A parent self-administered questionnaire including a parent's cognitive abilities test (self-administered);
3. Biological samples from the child (blood, urine, saliva hair)

ELIGIBILITY:
Inclusion Criteria:

* Children initially included in the Epipage 2 study,
* Not lost to follow up (i.e. having participated in at least one of the Epipage 2 surveys since the age of 1 year),
* Neither parent has expressed a definitive refusal to participate in the follow-up study.

Exclusion Criteria:

* Refusal of the investigation by one of the two parents or holders of parental authority,
* Residence abroad

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born before 35 weeks of amenorrhea still eligible for follow-up at 10 years of age
Sampling Method: Non-Probability Sample
Enrollment: 2383 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Relationships between prematurity, early growth and cardiometabolic disorders | 10 years and a half
  Different cardiometabolic parameters will be studied (90th percentile waist for age and sex, 90th percentile systolic or diastolic pressure for age and sex)
Relationship between parenting educational skills and children's quality of life | 10 years and a half
  VSPA scale (Adolescent Experience and Perceived Health)
Factors influencing children's puberty development | 10 years and a half
  Tanner stage
Factors influencing the child's fitness and motor skills | 10 years and a half
  Children's Endurance and Motor Ability Test Results upper or equal to 75th percentile of distribution for sex

CONTACTS AND LOCATIONS:
Locations (1):
- INSERM (National Institute of Health and Medical Research) - Université Paris Cité, INRAE, Obstetrical, Perinatal and Pediatric Epidemiology Research Team (EPOPé Team) Center for Epidemiology and Statistics, Paris, France

IPD SHARING:
Plan to Share IPD: No